CLINICAL TRIAL: NCT03172806
Title: Comparison of the New Algorithm of STOP-Bang in the Detection of Severe OSA Patients
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Investigator, Astes
Other Study IDs: NASB
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Apnea, Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: All patients included in the study. First: clinical scores were collected in all patients. Second: all patients underwent a polysomnography in order to compare this results with these of the clinical scores.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — To compare the ability of the clinical scores, all patients included in this study underwent a polysomnography.

SUMMARY:
The aim of this study was to compare the ability of clinical scores (P-SAP, OSA50, DES-OSA, STOP-Bang with former algorithm, and STOP-Bang with new algorithm).

DETAILED DESCRIPTION:
Severe OSA (Obstructive Sleep Apnea) patients are at higher risk of postoperative complications.

STOP-Bang has been proposed to detect OSA patients. It has been validated. New algorithm of STOP-Bang was proposed by the end of 2016. This aim of this study was to evaluate the ability of this new algorithm to detect severe OSA patients (patients with more than 30 events per hour). The new algorithm was also compared in this same ability with three others clinical score (P-SAP, OSA50 and DES-OSA).

ELIGIBILITY:
Inclusion Criteria:

* All patients in the preoperative anesthesia visit between 01/08/2016 and 31/12/2017

Exclusion Criteria:

* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolling in the preanesthsia visit before elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Comparison of results of clinical scores and results of polysomnography. | 1 night
  Comparison of the two results to determine the sensitivity and specificity of each clinical scores in comparison with polysmnography (the gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEFLANDRE, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc de Bouge, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No